CLINICAL TRIAL: NCT05911399
Title: Expanded Access Program for Tiratricol in Patients With Monocarboxylate Transporter 8 Deficiency Also Known as Allan-Herndon-Dudley Syndrome (AHDS)
Brief Title: Expanded Access Program for Tiratricol in Patients With Monocarboxylate Transporter 8 Deficiency
Status: Available | Type: Expanded Access
Sponsor: Rare Thyroid Therapeutics International AB (Industry)
Collaborators: AnovoRx (Unknown); Egetis Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: Tiratricol-EAP-Pro MCT8-2022-4
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Monocarboxylate Transporter 8 Deficiency; Allan-Herndon-Dudley Syndrome
Keywords: MCT8 Deficiency; Allan-Herndon-Dudley syndrome; Tiratricol; Triac; Expanded Access Program
MeSH Terms: conditions — Allan-Herndon-Dudley syndrome | interventions — 3,3',5-triiodothyroacetic acid

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Tiratricol — Tiratricol (3,3',5-triiodothyroacetic acid) is available as 350 µg tablets for oral administration (suspended in water and, if needed, mixed with food) or by percutaneous endoscopic gastrostomy (PEG), nasogastric or jejunal tube.

SUMMARY:
The goal of this program is to provide expanded access (i.e., before marketing authorization) to tiratricol as treatment for patients with monocarboxylate transporter 8 deficiency (MCT8 deficiency, also known as Allan-Herndon-Dudley syndrome [AHDS]), who in their Treating Physician's opinion, could benefit from tiratricol and meet the eligibility criteria.

DETAILED DESCRIPTION:
This will be an open-label, single-arm, multi-center EAP, designed to provide treatment access in the US to tiratricol for eligible patients with MCT8 deficiency, also known as AHDS.

Patients will undergo clinical and safety assessments before tiratricol treatment initiation, during the titration phase and then at approximately 3-6 monthly intervals or more frequently if clinically indicated, following the initiation of tiratricol treatment and until treatment is completed or discontinued.

Adverse events (AEs) and serious adverse events (SAEs) will be recorded and reported as per FDA regulations.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be eligible:

1. Diagnosis of MCT8 deficiency confirmed with a genetic test.
2. Either tiratricol treatment naïve, or patients who may be on a stable dose of tiratricol having transferred from the Phase 3 MCT8-2021-3 (ReTRIACt) study (NCT05579327) or prior individual investigational new drug (IND).
3. In the Treating Physician's medical opinion, the potential benefits of treatment with tiratricol outweigh the potential risks for the patient.
4. Patient or legal representative provided signed and dated informed consent to be treated with tiratricol, through this EAP.
5. Given the severity of the disease, sexual activity in these patients is deemed unlikely. However, where, at the discretion of the Treating Physician sexual activity is possible for the patient, patients must follow protocol-specified-contraception guidance.
6. Patient is approved for enrolment by the sponsor RTT.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the EAP:

1. Parents, legal representative or, if applicable, patients unwilling or unable to comply with the Treating Physician's treatment plan related to this EAP for any reason.
2. Major illness or recent major surgery unrelated to MCT8 deficiency (in the Treating Physician's judgement), defined as:

   * Conditions requiring repeated hospitalizations that are likely to confound ability to participate in the program.
   * Major illness in the 3 months before the screening visit that is likely to confound the ability of the patient to participate fully within the program and/or confound the assessment of serum total T3 and/or safety.
   * Major surgery within the 3 months before the screening visit, or planned to take place during the program, including but not limited to major abdominal/thoracic/neurosurgical procedures.
   * Major/minor abdominal and/or maxillofacial surgery that may inhibit the administration and/or absorption of tiratricol.
3. Patients with any contra-indication for treatment with tiratricol or any excipients in the program treatment.
4. Patients using thyroid hormone analogues- such as levothyroxine -or thionamides, such as propylthiouracil. Prior use of these drugs is not an exclusion criterion, provided the use of the medication has subsided and the thyroid hormone levels have stabilized after the cessation of these medications. For patients currently using these medications the switch to tiratricol should be made following the above and under the guidance of an endocrinologist with knowledge of MCT8 deficiency, if needed, after consultation with pharmacologist.
5. Known hypersensitivity to tiratricol including any ingredient in the pharmaceutical formulation.
6. Although very unlikely, as this is a severe X-linked disease: Women who are nursing or pregnant (or women who are planning to become pregnant during treatment with tiratricol).
7. Patients eligible for clinical trials with tiratricol.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Valley Children's Hospital - Enrollment limited to patients within the hospital's health system, Madera, California
  - Rady Children's Hospital, San Diego, California
  - Nemour's Children Hospital, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Louisiana State University Health Sciences Center and Children's Hospital, New Orleans, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - Gillette's Children's Specialty Healthcare, Saint Paul, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital Foundation, Memphis, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - MultiCare Mary Bridge Children's Hospital, Tacoma, Washington
  - Children's Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Groeneweg S, Peeters RP, Moran C, Stoupa A, Auriol F, Tonduti D, Dica A, Paone L, Rozenkova K, Malikova J, van der Walt A, de Coo IFM, McGowan A, Lyons G, Aarsen FK, Barca D, van Beynum IM, van der Knoop MM, Jansen J, Manshande M, Lunsing RJ, Nowak S, den Uil CA, Zillikens MC, Visser FE, Vrijmoeth P, de Wit MCY, Wolf NI, Zandstra A, Ambegaonkar G, Singh Y, de Rijke YB, Medici M, Bertini ES, Depoorter S, Lebl J, Cappa M, De Meirleir L, Krude H, Craiu D, Zibordi F, Oliver Petit I, Polak M, Chatterjee K, Visser TJ, Visser WE. Effectiveness and safety of the tri-iodothyronine analogue Triac in children and adults with MCT8 deficiency: an international, single-arm, open-label, phase 2 trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):695-706. doi: 10.1016/S2213-8587(19)30155-X. Epub 2019 Jul 31. PMID 31377265
- [Background] van Geest FS, Groeneweg S, van den Akker ELT, Bacos I, Barca D, van den Berg SAA, Bertini E, Brunner D, Brunetti-Pierri N, Cappa M, Cappuccio G, Chatterjee K, Chesover AD, Christian P, Coutant R, Craiu D, Crock P, Dewey C, Dica A, Dimitri P, Dubey R, Enderli A, Fairchild J, Gallichan J, Garibaldi LR, George B, Hackenberg A, Heinrich B, Huynh T, Klosowska A, Lawson-Yuen A, Linder-Lucht M, Lyons G, Monti Lora F, Moran C, Muller KE, Paone L, Paul PG, Polak M, Porta F, Reinauer C, de Rijke YB, Seckold R, Menevse TS, Simm P, Simon A, Spada M, Stoupa A, Szeifert L, Tonduti D, van Toor H, Turan S, Vanderniet J, de Waart M, van der Wal R, van der Walt A, van Wermeskerken AM, Wierzba J, Zibordi F, Zung A, Peeters RP, Visser WE. Long-Term Efficacy of T3 Analogue Triac in Children and Adults With MCT8 Deficiency: A Real-Life Retrospective Cohort Study. J Clin Endocrinol Metab. 2022 Feb 17;107(3):e1136-e1147. doi: 10.1210/clinem/dgab750. PMID 34679181